CLINICAL TRIAL: NCT01518543
Title: Follow-up of Patient Implanted With the Staple ASTUS®
Status: Terminated | Type: Observational
Sponsor: Integra LifeSciences Services (Industry)
Responsible Party: Sponsor
Other Study IDs: RECON-EMEA-04
Record Dates: First submitted 2011-06-20; First posted 2012-01-26 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Arthrodesis
Keywords: arthrodesis; arthrodesis in the following joints:Ankle, 1st MTP, Metatarso - Cuneiform (1st), Navicular - Cuneiform, Talo-Navicular, Calcaneum - Cuboid;
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ASTUS: Patient candidate for an arthrodesis in the following joints:Ankle,1st MTP, Metatarso - Cuneiform (1st), Navicular - Cuneiform, Talo-Navicular, Calcaneum - Cuboid, and whose surgeon has recommended the implantation of an ASTUS Staple from Newdeal-INTEGRA.

SUMMARY:
There are many ways of performing arthrodesis in the foot and ankle. Dowel fusion is one of them.

The in situ technique was first described by Ottolenghi et al. (1970) and was taken up by Baciu and Filibiu (1979). In the technique, they did take the dowel out before turning it. The healing process takes place between surfaces of spongious bone. They showed excellent results with early weight bearing and healing within 12.5 weeks. Stranks et al. (1994) combined the dowel technique with screw fixation and claimed 95 % healing rate within 12.5 weeks. Others have not found this technique satisfactory in rheumatoid arthritis patients (Belt et al. 2001). The results were not compatible to common fusion techniques. The reason may be the circular bone gap of at least 1 mm left by the saw blade.

A new instrumentation and a new staple with a central wedge (ASTUS) avoid this gap and allow the dowel to be turned in situ without leaving in position. The staple is introduced into the joint line and will compress the dowel surfaces against the surrounding bone. Instruments are available to ensure the correct position and length of the dowel, and to rotate it in situ before the special wedge staple is introduced.

Dr Kofoed, the surgeon designer of the ASTUS Staple, has communicated on his first series with 83 arthrodesis. The purpose of this study is now to collect and publish data from several centers, several users.

The objective of this study is to obtain the percentage of healing 3 months after an implantation of the staple ASTUS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Have willingness to give his/her data transfer authorisation;
* Patient candidate for an arthrodesis in the following joints (Ankle, 1st MTP, Metatarso - Cuneiform (1st), Navicular - Cuneiform, Talo-Navicular, calcaneum - Cuboid) and whose surgeon has recommended the implantation of an ASTUS Staple from Newdeal-INTEGRA.

Exclusion Criteria:

* Patient candidate for an arthrodesis not listed in the inclusion criteria (as Subtalar arthrodesis and Metatarso-cuboid arthrodesis) will not be included in this study;
* Patient re-operated due to a previous failed of fusion of the same joint will not be also included;
* Patients will be excluded from the study if they have an history of prior mental illness or patient demonstrates that their mental capacity may interfere with their ability to follow the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient candidate for an arthrodesis in the following joints (Ankle, 1st MTP, Metatarso - Cuneiform (1st), Navicular - Cuneiform, Talo-Navicular, calcaneum - Cuboid) and whose surgeon has recommended the implantation of an ASTUS Staple from Newdeal-INTEGRA can be enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Rate of healing at 3 month | 3 month post implantation

SECONDARY OUTCOMES:
Complications rate | 12 month follow-up
  Number of patients with an adverse event related to the device
Length of the surgery | The time is the day of the surgery, the day the implantation of the device is done
  We collect the information of the length of the surgery for the implantation of the Astus Device

CONTACTS AND LOCATIONS:
Locations (2):
- Cappagh National Orthopaedic Hospital, Dublin, Ireland
- Clatterbridge General Hospital, Metropolitan Borough of Wirral, United Kingdom